CLINICAL TRIAL: NCT01452386
Title: Modified Functional Magnetic Stimulation Treatment for Constipation Improvement
Status: Withdrawn | Type: Observational
Why Stopped: no sufficient subjects
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Fat-Moon Suk, Principal Investigator, Taipei Medical University WanFang Hospital
Other Study IDs: 99081
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Constipation
Keywords: Constipation; Stimulation Treatment
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
To prove the modify functional magnetic stimulation could improve constipation.

DETAILED DESCRIPTION:
1. Permission： Any agent without effecting gastrointestinal motility or defecation is allowed.
2. Inhibition： From test day to the next day(48 hours),it's not allowed to take any medication treatment which might affect digestive system or excretory system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who age between 20~60 years old and have suffered from chronic constipation for more than 6 months will be enrolled in this study.

Exclusion Criteria:

* Patients with implantation chip of brain
* Patients with implantation of pacemaker
* Patients with heart transplantation
* Patients are embedded electronic and Life support products.
* People who have be implanted metal、electronic devices、artificial joints or fixator.
* Patients with hemiplegia
* Patients with peripheral neuritis
* Patients with Prostate abnormalities
* Patients with Pregnancy
* Patients with Fever
* Patients with Injure
* Patients with Heart disease
* Patients with Consciousness disturbance
* Patients with Organic constipation
* Patients with Kidney stone
* Patients with Ureteric calculus

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: constipation patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
To improve bowel movement by the modify functional magnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Fat-Moon Suk, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan